CLINICAL TRIAL: NCT03691337
Title: Fascia Iliaca Block for Analgesia in Unilateral Direct Anterior Approach Total Hip Arthroplasty
Brief Title: Fascia Iliaca Blocks for Total Hip Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: New York School of Regional Anesthesia (Other)
Responsible Party: Principal Investigator, Catherine Vandepitte, M.D., Medical Doctor, New York School of Regional Anesthesia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1802
Record Dates: First submitted 2018-08-01; First posted 2018-10-01 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: THA
MeSH Terms: interventions — Bupivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low dosis bupivacaine (Active Comparator): Preoperative fascia iliaca block with Marcaine 0.25% (0.11 mL x subject height)
  Interventions: Drug: Marcaine 0.25 % Injectable Solution
- High dosis bupivacaine (Active Comparator): Preoperative fascia iliaca block with Marcaine 0.25% (0.22 mL x subject height)
  Interventions: Drug: Marcaine 0.25 % Injectable Solution
- Placebo (Placebo Comparator): Preoperative fascia iliaca block with Sodium Chloride 0.9% (0.11 mL x subject height)
  Interventions: Drug: Sodium chloride

INTERVENTIONS:
Drug: Marcaine 0.25 % Injectable Solution — Fascia iliaca block with volume 0.11 mL x subject height
  Arms: Low dosis bupivacaine
Drug: Marcaine 0.25 % Injectable Solution — Fascia iliaca block with volume 0.22 mL x subject height
  Arms: High dosis bupivacaine
Drug: Sodium chloride — Fascia iliaca block with volume 0.11 mL x subject height
  Arms: Placebo

SUMMARY:
The development of minimal-incision techniques for total hip arthroplasty (THA) with preservation of soft tissue is generally associated with reduction of postoperative pain and increased patient comfort. Although this technique requires a smaller incision than other approaches used for hip surgery, adequate postoperative pain management remains crucial for enhanced recovery and early rehabilitation. The fascia iliaca block (FIB) is commonly used to enhance analgesia after hip replacement surgery, however the effect of FIB volume on analgesia quality and sensory-motor blockade have not been adequately studied. In this study, total postsurgical opioid consumption (morphine equivalents IV in hospital and oral at home) through the first postoperative week will be compared and extent and duration of sensory motor block through the 2-day inpatient stay will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, at least 18 years of age at screening
* Scheduled for unilateral DAA THA
* American Society of Anesthesiologists (ASA) physical status 1, 2 or 3
* Able to demonstrate sensory function by exhibiting sensitivity to light touch, pinprick and cold
* Able to ambulate
* Able to provide informed consent, adhere to the study visit schedule, and complete all study assessments

Exclusion Criteria:

* Previous open hip surgery
* History of hypersensitivity or idiosyncratic reaction to amide-type local anesthetics
* Contraindication to bupivacaine or morphine
* Concurrent physical condition that may require analgesic treatment (such as NSAID or opioid) in the postsurgical period for pain that is not strictly related to the hip surgery and which may confound the postsurgical assessments
* Initiation of treatment with any of the following medications within 1 month of study drug administration or if the medication(s) are being given to control pain: selective serotonin reuptake inhibitors (SSRIs), selective norepinephrine reuptake inhibitors (SNRIs), gabapentin, pregabalin (Lyrica®), or duloxetine (Cymbalta®)
* Body weight <40 kg (88 pounds) or a body mass index >44 kg/m2
* Uncontrolled anxiety, psychiatric, or neurological disorder that might interfere with study assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2018-05-15 (Actual); Primary Completion 2019-11-12 (Actual); Study Completion 2019-12-04 (Actual)

PRIMARY OUTCOMES:
Current pain assessed by numeric rating scale (NRS) | Day 0
  Pain rating (Numeric Rating Scale: 0 (no pain) - 10 (worst pain)) at rest and with movement
Current pain assessed by numeric rating scale (NRS) | PACU arrival
  Pain rating (Numeric Rating Scale: 0 (no pain) - 10 (worst pain)) at rest and with
Current pain assessed by numeric rating scale (NRS) | PACU discharge
  Pain rating (Numeric Rating Scale: 0 (no pain) - 10 (worst pain)) at rest and with
Current pain assessed by numeric rating scale (NRS) | 6 hours
  Pain rating (Numeric Rating Scale: 0 (no pain) - 10 (worst pain)) at rest and with
Current pain assessed by numeric rating scale (NRS) | 12 hours
  Pain rating (Numeric Rating Scale: 0 (no pain) - 10 (worst pain)) at rest and with
Current pain assessed by numeric rating scale (NRS) | 24 hours
  Pain rating (Numeric Rating Scale: 0 (no pain) - 10 (worst pain)) at rest and with
Current pain assessed by numeric rating scale (NRS) | 36 hours
  Pain rating (Numeric Rating Scale: 0 (no pain) - 10 (worst pain)) at rest and with
Current pain assessed by numeric rating scale (NRS) | 48 hours
  Pain rating (Numeric Rating Scale: 0 (no pain) - 10 (worst pain)) at rest and with
Current pain assessed by numeric rating scale (NRS) | Day 2 evening
  Pain rating (Numeric Rating Scale: 0 (no pain) - 10 (worst pain)) at rest and with
Current pain assessed by numeric rating scale (NRS) | Day 3 morning
  Pain rating (Numeric Rating Scale: 0 (no pain) - 10 (worst pain)) at rest and with
Current pain assessed by numeric rating scale (NRS) | Day 3 evening
  Pain rating (Numeric Rating Scale: 0 (no pain) - 10 (worst pain)) at rest and with
Current pain assessed by numeric rating scale (NRS) | Day 4
  Pain rating (Numeric Rating Scale: 0 (no pain) - 10 (worst pain)) at rest and with
Current pain assessed by numeric rating scale (NRS) | Day 5
  Pain rating (Numeric Rating Scale: 0 (no pain) - 10 (worst pain)) at rest and with
Current pain assessed by numeric rating scale (NRS) | Day 6
  Pain rating (Numeric Rating Scale: 0 (no pain) - 10 (worst pain)) at rest and with
Current pain assessed by numeric rating scale (NRS) | Day 7
  Pain rating (Numeric Rating Scale: 0 (no pain) - 10 (worst pain)) at rest and with

SECONDARY OUTCOMES:
Total opioid consumption | PACU arrival
  Amount of opioid medication taken (IVPCA or oral)
Total opioid consumption | PACU discharge
  Amount of opioid medication taken (IVPCA or oral)
Total opioid consumption | 6 hours
  Amount of opioid medication taken (IVPCA or oral)
Total opioid consumption | 12 hours
  Amount of opioid medication taken (IVPCA or oral)
Total opioid consumption | 24 hours
  Amount of opioid medication taken (IVPCA or oral)
Total opioid consumption | 36 hours
  Amount of opioid medication taken (IVPCA or oral)
Total opioid consumption | 48 hours
  Amount of opioid medication taken (IVPCA or oral)
Total opioid consumption | Day 2 evening
  Amount of opioid medication taken (IVPCA or oral)
Total opioid consumption | Day 3 morning
  Amount of opioid medication taken (IVPCA or oral)
Total opioid consumption | Day 3 evening
  Amount of opioid medication taken (IVPCA or oral)
Total opioid consumption | Day 4
  Amount of opioid medication taken (IVPCA or oral)
Total opioid consumption | Day 5
  Amount of opioid medication taken (IVPCA or oral)
Total opioid consumption | Day 6
  Amount of opioid medication taken (IVPCA or oral)
Total opioid consumption | Day 7
  Amount of opioid medication taken (IVPCA or oral)
Sensory-motor blockade onset and duration | Day 0
  Cold, pinprick, light touch in affected dermatomes + strength and angle of knee
Sensory-motor blockade onset and duration | Post block
  Cold, pinprick, light touch in affected dermatomes + strength and angle of knee
Sensory-motor blockade onset and duration | PACU arrival
  Cold, pinprick, light touch in affected dermatomes + strength and angle of knee
Sensory-motor blockade onset and duration | PACU discharge
  Cold, pinprick, light touch in affected dermatomes + strength and angle of knee
Sensory-motor blockade onset and duration | 6 hours
  Cold, pinprick, light touch in affected dermatomes + strength and angle of knee
Sensory-motor blockade onset and duration | 12 hours
  Cold, pinprick, light touch in affected dermatomes + strength and angle of knee
Sensory-motor blockade onset and duration | 36 hours
  Cold, pinprick, light touch in affected dermatomes + strength and angle of knee
Sensory-motor blockade onset and duration | 48 hours
  Cold, pinprick, light touch in affected dermatomes + strength and angle of knee

CONTACTS AND LOCATIONS:
Locations (1):
- Ziekenhuis Oost-Limburg, Genk, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: Undecided